CLINICAL TRIAL: NCT04908267
Title: To Determine Whether the Habitats Created by the Preoperative or Postoperative Multiparametric MRI Can Predict IDH Mutation Status, Prognosis, Recurrence or Intracranial Distant Recurrence of the Patients With High-grade Gliomas
Brief Title: How the Precise Habitats Can Predict the IDH Mutation Status and Prognosis of the Patients With High-grade Gliomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weiguo Zhang (Other)
Responsible Party: Sponsor-Investigator, Weiguo Zhang, Director of Radiology Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: 2022198
Record Dates: First submitted 2021-05-17; First posted 2021-06-01 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: High-grade Glioma
Keywords: habitat imaging; high-grade glioma; radiomics; heterogeneity; recurrence
MeSH Terms: conditions — Glioma; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High-grade glioma is the most common primary malignant tumor in central nervous system, and its high tumor heterogeneity is the main cause of tumor progression, treatment resistance and recurrence. Habitat imaging is a segmentation technique by dividing tumor regions to characterize tumor heterogeneity based on tumor pathology, blood perfusion, molecular characteristics and other tumor biological features.

In some studies, the Hemodynamic Multiparametric Tissue Signature (HTS) method has been proven to be feasible. The Hemodynamic Multiparametric Tissue Signature (HTS) consists of a set of vascular habitats obtained by Dynamic Susceptibility Weighted Contrast Enhanced Magnetic Resonance Imaging (DSC-MRI) of high-grade gliomas using a multiparametric unsupervised analysis method. This allowed them to automatically draw 4 reproducible vascular habitats (High-angiogenic enhancing tumor; Low-angiogenic enhancing tumor; Potentially tumor infiltrated peripheral edema; Vasogenic peripheral edema) which enable to describe the tumor vascular heterogeneity robustly.

In other studies, contrast-enhancing mass can divided into spatial habitats by K-means clustering of voxel-wise apparent diffusion coefficient (ADC) and cerebral blood volume (CBV) values to observe the changes of voxels in spatial habitat on the time line. Using this so-called spatiotemporal habitat to identify progression or pseudoprogression in cancer therapy.

Above all, we have sufficient and firm reasons to deem that habitat imaging based on multiparametric MRI is more conducive to reflect the potential biological information inside the tumor and realize individualized diagnosis and treatment.

To sum up, the assumption of this experiment is that the Habitats Created by preoperative or postoperative Multiparametric MRI ,such as conventional MRI sequences, Dynamic Susceptibility Weighted Contrast Enhanced Magnetic Resonance Imaging (DSC-MRI), Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE-MRI), Diffusion Weighted Magnetic Resonance Imaging(DWI) ,Vessel Size Imaging (VSI) ,or Magnetic Resonance Spectroscopy (MRS) can predict the molecular mutation status, prognosis, treatment residence, progression, pseudoprogression, and even recurrence and distant intracranial recurrence in patients with high-grade gliomas.

DETAILED DESCRIPTION:
This is a single center experiment. The subjects of this study were patients diagnosed as high-grade glioma by multiparametric magnetic resonance imaging and pathological biopsy from January 1, 2008 to December 31, 2021(or at some interval within this period). Patients meeting the inclusion criteria will enter the next experimental stage.

1. Patients selection: The patients will be clustered according to the preoperative and postoperative examination methods performed by each patient, such as only DSC sequence, both DSC and DWI sequences, or a full set of functional imaging sequences at the same time;
2. Images segmentation: To select the patients who meet the experimental design, and use deep learning-based biomedical image segmentation methods, such as Brain Tumor Segmentation (BraTS) challenge, to segment more accurate and reproducible habitats as much as possible;
3. Construction of clinical model: We may be able to obtain the parameter values of the habitat, such as CBV, ADC, Ktrans, etc. Combining these data with the basic situation of patients can build a clinical model.
4. Construction of radiomics model: The radiomics analysis will probably be structured into four parts: habitats segmentation, feature extraction, feature selection and model construction.
5. We try to analyze that habitat imaging based on Multiparametric MRI is indeed better than the conventional rough and simple ROI analysis; We try to analyze the relation between the habitats and the IDH mutation status or MGMT promoter methylation status; We try to analyze the relation between the habitats and the overall survival (OS) of the patient; We try to analyze the habitats is conducive to differentiate recurrence from distant intracranial recurrence.

Finally, statistical methods and survival analysis were used to determine whether the habitat was statistically significant for IDH mutation status and prognosis. For example, receiver operating characteristic curve (ROC) analysis evaluated the potential of the spatial habitats in IDH mutation prediction. The Kaplan-Meier curve evaluates the validation of the diagnosis in OS prediction in high-grade glioma.

ELIGIBILITY:
Inclusion Criteria (if we will predict the molecular status and overall survival):

* the patient was over 18 years old
* the lesion was located in the supratentorial space;
* a histopathologic diagnosis of HGGs according to the WHO CNS4/5;
* all subjects were the first diagnosed cases without any invasive or non-invasive treatment;
* access to the complete preoperative MR imaging examinations, at least including four conventional sequences.

Inclusion Criteria (if we will differentiate recurrence from distant intracranial recurrence):

* the patient was over 18 years old;
* the lesion was located in the supratentorial space;
* a histopathologic diagnosis of HGGs according to the WHO CNS4/5;
* underwent concurrent chemoradiotherapy with temozolomide after surgical resection or biopsy;
* underwent preoperative and postoperative MRI, at least including four conventional sequences;
* had newly appeared or enlarging, measurable, contrast-enhancing mass which raises clinical suspicion of tumor recurrence and distant intracranial recurrence;
* adequate follow-up examinations to determine treatment response on clinic-radiological consensus or pathologic confirmation.

Exclusion Criteria:

* patient with other brain tumors or other grade gliomas at the same time;
* patient with severe basic diseases at the same time;
* patient with a survival time of less than 30 days, which can be caused by severe surgical trauma stress;
* poor image quality and heavy artifact affect the subsequent image processing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects we selected are adults who are not restricted by gender. For details, please refer to the "criteria" column.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Multi-model habitats constructed by multiparametric MRI predict IDH mutation status and the prognosis in high-grade gliomas | From the date of operation until the date of death from any cause，assessed up to 120 months
  The IDH status of each patient was dependent on pathological and immunohistochemical results. The overall survival for each patient is estimated since the date of operation to the end of recruitment. The overall survival will be confirmed through clinical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Zhang, Ph.D, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of Radiology, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu H, Tong H, Du X, Guo H, Ma Q, Zhang Y, Zhou X, Liu H, Wang S, Fang J, Zhang W. Vascular habitat analysis based on dynamic susceptibility contrast perfusion MRI predicts IDH mutation status and prognosis in high-grade gliomas. Eur Radiol. 2020 Jun;30(6):3254-3265. doi: 10.1007/s00330-020-06702-2. Epub 2020 Feb 20. PMID 32078014
- See also: Vascular habitat analysis based on dynamic susceptibility contrast perfusion MRI predicts IDH mutation status and prognosis in high-grade gliomas — http://pubmed.ncbi.nlm.nih.gov/32078014/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04908267/Prot_SAP_000.pdf